CLINICAL TRIAL: NCT06216548
Title: Enhanced Primary Care Via Telehealth for Children With Medical Complexity
Brief Title: E-PRIME For Children With Medical Complexity
Acronym: E-PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00102234; TE-2022C3-30607 (Other: PCORI)
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Children With Medical Complexity
Keywords: Collaboration; Providers; Telehealth

STUDY DESIGN:
Intervention Model Description: Intervention participants will complete the Enhanced Primary Care via Telehealth (E-PRIME) intervention for 12 months while Comparison participants will receive usual care for 6 months then complete the E-PRIME intervention for 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Enhanced Primary Care (E-PRIME) Group (Active Comparator): Children will receive usual care before receiving E-PRIME intervention.
  Interventions: Other: Usual Care and Enhanced Primary Care
- Early Enhanced Primary Care (E-PRIME) Group (Experimental): Subjects of this arm will receive E-PRIME intervention at the start of enrollment.
  Interventions: Other: Enhanced Primary Care

INTERVENTIONS:
Other: Usual Care and Enhanced Primary Care — Usual Care: Interdisciplinary complex care teams help coordinate appointments, facilitate communication between the many specialist providers involved in the child's care, support families, assist with practical needs, and are available as a resource (as consultants) for Primary Care Physicians (PCPs) to care for Children with Medical Complexity (CMC). The complex care teams in tertiary care children's hospital is the focus for providing comprehensive care for CMC.
  Enhanced Primary Care: The E-PRIME team will support the CMC and their caregivers with navigating the patient access portal and how to use the video visit platform for the telehealth visits. The physician or nurse of the E-PRIME team will create clinical summaries about CMC's visit to specialists and hospital and share this health information about CMC with his/her PCP to help the PCP provide care for CMC at home. A team of telehealth experts will help PCPs in using telehealth in their practice.
  Other Names: Delayed E-PRIME
  Arms: Delayed Enhanced Primary Care (E-PRIME) Group
Other: Enhanced Primary Care — The intervention has the following components: (A) The staff of the E-PRIME team will support the CMC and their caregivers with navigating the patient access portal and how to use the video visit platform for the telehealth visits. (B) The physician or nurse of the E-PRIME team will create clinical summaries about CMC's visit to specialists and hospital and share this health information about CMC with his/her PCP to help the PCP provide care for CMC at home. (C) A team of telehealth experts will help PCPs in using telehealth in their practice.
  Other Names: E-PRIME
  Arms: Early Enhanced Primary Care (E-PRIME) Group

SUMMARY:
Children with medical complexity (CMC) have very high needs for health and support services. CMC have very rare diseases that involve multiple organ systems. As a result, all CMC have multiple chronic conditions and need care from many specialists and services. While there are important benefits to the child and family in living at home, the continuing need for complex medical care places a profound burden on caregivers. Telehealth has long been considered a potential solution to barriers in access to care for children. The purpose of this research is to test whether telehealth can help pediatric primary care providers (PCPs) as they treat, monitor, and manage children with medical complexity (CMC). Additionally, it is to reduce caregiver and child burden as well as improve care coordination between multiple providers.

DETAILED DESCRIPTION:
The specific aims of this study are to: compare the effectiveness of Enhanced Primary Care via Telehealth (E-PRIME) verses usual care in improving child-level appointment and outcome measures; compare the effectiveness of (E-PRIME) verses usual care in reducing caregiver stress and improving caregiver satisfaction in primary care and care coordination services; evaluate how acceptable, appropriate, and feasible E-PRIME is from the perspective of practice providers and staff, and caregivers. Telehealth has long been considered a potential solution to barriers in access to care for children. The purpose of this research is to test whether telehealth can help pediatric primary care providers (PCPs) as they treat, monitor, and manage children with medical complexity (CMC). Additionally, it is to reduce caregiver and child burden as well as improve care coordination between multiple providers.

ELIGIBILITY:
Inclusion Criteria:

* Less than 18 years of age on the date of enrollment (date consented)
* Presence of a chronic condition, defined as a health condition expected to last ≥ 12 months
* Complexity of the condition, defined as needing ongoing care with 4 sub-specialists/ services OR dependent on ≥ 1 technology (e.g. gastrostomy, tracheostomy, oxygen, ventilator, etc.)

Exclusion Criteria:

* CMC whose permanent address is outside of the state of North Carolina
* CMC at a long-term care facility
* CMC who are wards of the state, except when the caregiver is a legal guardian and can consent
* CMC whose caregivers do not speak English or Spanish

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 909 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Number of Days Outside the Home (DOH) | Baseline
  Number of hospital days + ER visit days + number of in-person appointments / child year
Number of Days Outside the Home (DOH) | Year 1
  Number of hospital days + ER visit days + number of in-person appointments / child year

SECONDARY OUTCOMES:
Number of Hospitalizations | Year 1
  Number of hospitalizations/100-child years in the two groups. Number of hospitalizations during the observation period will be counted and the rate will be calculated as: [Number of hospitalizations/ observation period in years]*100. Planned admissions (i.e. elective surgeries, procedures, treatments, etc.) will be excluded.
Number of Emergency Room (ER) visits | Year 1
  Number of ER visits
Number of Hospital Days | Year 1
  Number of hospital days/observation period in years
Appointment Completion Rate | Year 1
  Proportion of scheduled appointments that were completed
Change in Caregiver Burden scores | Month 19
  Caregiver burden will be measured using the 15-item Impact on Family Scale- Revised which as 15 items and 4 domains - financial, family/social, personal strain, and mastery. Scores will range from 15 to 60. The higher the score the greater the impact.
Change in Caregiver Satisfaction with coordination of care scores | Month 19
  Caregiver satisfaction with coordination of care will be compared between the two groups and measured by the Family Experiences with Coordination of Care survey. Scores will range from 0 to 100 and each item will be measured independently. Higher scores indicate better care (i.e. care plans, coordination, visit summary content, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Savithri Nageswaran, MD, Principal Investigator — Wake Forest University Health Sciences; Sabina Gesell, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No